CLINICAL TRIAL: NCT04069169
Title: Perioperative Multimodal Analgesia Including Intravenous Lidocaine Infusion for Pain Management Following Idiopathic Scoliosis Correction Surgery in Children
Brief Title: IV Lidocaine Analgesia in Pediatric Scoliosis Surgery
Acronym: P-IVLT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Gillian Lauder, Staff Anesthesiologist, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: H18-03103
Record Dates: First submitted 2019-05-13; First posted 2019-08-28 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Scoliosis; Adolescence; Anesthesia Recovery Period
MeSH Terms: conditions — Scoliosis | interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Intervention Model Description: This will be a placebo-controlled, double-blind randomized control trial (RCT) comparing 48-hour postoperative morphine utilization amongst adolescents undergoing posterior spinal instrumentation and fusion who have been randomly assigned to one of two groups:
  1. Intervention group will receive perioperative IV lidocaine therapy (1% preservative free lidocaine 10 mg/ml in 0.9% NaCl) in addition to the standard multi-modal analgesia.
  2. Control group will receive a placebo (0.9% sodium chloride also known as normal saline), made to mimic the intervention.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Following receipt of informed consent, participants will be randomized by the Pharmacy Research Support Pharmacist. Pharmacy research staff will prepare an appropriate randomization schedule (patients randomized to P-IVLT or control) and deploy blinded study drug to the operating room, anesthesia care unit, and post-surgical ward as required. Unless emergency unblinding is required, the following people will remain blinded to group allocation until the full cohort has been recruited and data collection has been completed:
  1. All anesthesia, APS, nursing, clinical pharmacists and surgical staff involved in the patient's clinical care
  2. The patient and their family
  3. Research staff involved in recruitment and data collection
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intravenous lidocaine (Experimental): 1% preservative free lidocaine 10 mg/ml in 0.9% NaCl
  Interventions: Drug: Lidocaine
- Intravenous saline control (Placebo Comparator): 0.9% sodium chloride, also known as normal saline
  Interventions: Drug: Saline Solution

INTERVENTIONS:
Drug: Lidocaine — Intervention group (A) will receive P-IVLT in addition to the standard multimodal analgesia. P-IVLT will consist of 1 mg/kg bolus at start of anesthesia (T0), followed by 2 mg·kg-1·hr-1 infusion for 8 hours (T1), then continued at 1 mg·kg-1·hr-1 infusion thereafter and postoperatively until T0 + 48 hours (T2).
  Arms: Intravenous lidocaine
Drug: Saline Solution — Control group (B) will receive a placebo (0.9% sodium chloride also known as normal saline), made to mimic the intervention protocol described above, in addition to the standard multimodal analgesia.
  Arms: Intravenous saline control

SUMMARY:
Surgical correction of scoliosis in children is a long procedure, with an equivalently long recovery time, that is commonly performed at BC Children's Hospital. Treating pain immediately after the procedure is a priority for children during recovery. Morphine is one medication that can be used to manage post-operative pain, but unfortunately, its use is accompanied by a number of side effects which can affect recovery. These include nausea, vomiting, pruritus, sedation, dysphoria, respiratory depression, constipation, ileus, and urinary retention.

In order to control pain and reduce morphine consumption, intravenous lidocaine is being investigated. This therapy has been beneficial in adult populations undergoing abdominal surgery and has been associated with decreased post-operative pain, decrease use of opioids including morphine, and ileus. These all contribute to shorter lengths of stay in the hospital and better recovery in the adult population.

Intravenous lidocaine is used by some anesthesiologists at BC Children's Hospital to manage post-operative pain in children receiving surgical correction for scoliosis, but this is not a standard of practice. We now propose to conduct a double-blind randomized controlled trial to determine if intravenous lidocaine, infused from start of anesthesia up to 48 hours post-operatively, will reduce morphine use and improve post-operative pain in the pediatric population.

DETAILED DESCRIPTION:
Objectives:

The primary objective of this study is to determine if perioperative IV lidocaine therapy (P-IVLT) reduces 48-hour post-operative morphine utilization compared with a control, in adolescents undergoing PSIF. Secondary objectives of this study are to determine the effect of P-IVLT on self-reported pain scores, time to documented first stand, time to first walk of greater than 15 steps, and length of hospital stay (LOS).

Research Methods:

This will be a placebo-controlled, double-blind randomized control trial (RCT) comparing 48-hour postoperative morphine utilization among adolescents undergoing PSIF who have been randomly assigned to one of two groups:

Intervention group (A) will receive P-IVLT in addition to the standard multimodal analgesia. P-IVLT will consist of 1 mg/kg bolus at start of anesthesia (T0), followed by 2 mg·kg-1·hr-1 infusion for 8 hours (T1), then continued at 1 mg·kg-1·hr-1 infusion thereafter and postoperatively until T0 + 48 hours (T2).

Control group (B) will receive a placebo (0.9% sodium chloride also known as normal saline), made to mimic the intervention protocol above, in addition to the standard multimodal analgesia.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* Diagnosed with Idiopathic scoliosis
* Undergoing single-stage posterior spinal instrumentation and fusion

Exclusion Criteria:

* Thorascopic tethering procedure
* Two-stage procedure
* Abnormal developmental profile
* Congenital/neuromuscular scoliosis
* Requiring PICU admission
* Known allergy to lidocaine
* Known cardiac, renal or liver disease or dysfunction
* Pre-existing pain complaints, i.e. on regular analgesic medications
* Current psychiatric diagnosis, e.g. anxiety, depression, eating disorder, defined according to DSM criteria.
* Requiring non-standard post-op pain management
* Any history of seizures
* Unplanned staged procedure
* Weight < 5th centile or > 85th centile for age
* Porphyria

Ages: 10 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 48 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-05-10 (Actual)

PRIMARY OUTCOMES:
Total morphine utilization | 48 hours post-operatively
  Documented from acute pain service charts (mg/kg)

SECONDARY OUTCOMES:
Total morphine utilization | 12, 24, 36 hours post-operatively
  Documented from acute pain service charts (mg/kg)
Postoperative pain | from emergence in the anesthetic care unit through 48 hours post-operatively
  Pain scores measured every 4 hours by nursing staff
Mobililzation | through hospital stay, an average of 5 days
  Time from anesthesia induction to first walk of greater than 15 steps (hours)
Urinary incontinence | through hospital stay, an average of 5 days
  Time from anesthesia induction to urinary catheter removal (hours)
Postoperative pain (II) | through study completion, 48 hours post-operatively
  Time from anesthesia induction to termination of morphine (hours)
Recovery | through hospital stay, an average of 5 days
  Time from anesthesia induction to discharge from hospital (days)

CONTACTS AND LOCATIONS:
Overall Officials: Gill Lauder, MD, Principal Investigator — University of British Columbia
Locations (1):
- BC Children's Hospital - Department of Anesthesia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luo J, West N, Pang S, Golam A, Adams E, Gorges M, Carr RR, Miyanji F, Lauder GR. Perioperative Intravenous Lidocaine Infusion Therapy as an Adjunct to Multimodal Analgesia for Adolescent Idiopathic Scoliosis Surgical Correction: A Double-Blind Randomized Controlled Trial. Paediatr Anaesth. 2025 Jul;35(7):552-561. doi: 10.1111/pan.15124. Epub 2025 May 6. PMID 40326715
- See also: Pediatric Anesthesia Research Team website — http://bcchr.ca/PART